CLINICAL TRIAL: NCT04162561
Title: Trying to Improve Quality of therApy in Patients With stabLe Coronary Artery dIsease According to Current Clinical GuideliNes (ALIGN)
Brief Title: TherApy in stabLe Coronary Artery dIsease Patients According to Clinical GuideliNes (ALIGN)
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: PROFILE
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Stable Ischemic Heart Disease
Keywords: quality of therapy; current clinical guidelines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Patients with documented IHD — Assessment of patients' quality of life with the use of the Seattle Angina Questionnaire (SAQ), blood pressure levels (using the Korotkoff method, blood pressure is measured 3 times with 1-minute intervals on the hand with the higher blood pressure levels while sitting calm after a 5-minutes rest), laboratory methods (lipids, glycosylated hemoglobin levels), patients' adherence to treatment (original questionnaire), quality of patients' therapy taken at the time of visit, necessity of invasive coronary revascularization procedures (during all visits).

SUMMARY:
The aim of this prospective cohort study is to assess the quality of therapy in patients with stable ischemic heart disease (IHD) who had never applied for specialized medical care for the last 3 years and try to accord their treatment with current clinical guidelines.

DETAILED DESCRIPTION:
The purpose of this study is to assess the quality of therapy in patients having come for the first time consultation to the specialized cardiology department of the scientific research centre within the PROFILE registry and to try to correct therapy according to current clinical guidelines paying particular attention to reaching target blood pressure (BP), low-density lipoprotein cholesterol (LDL-C), glycosylated haemoglobin - HbA1c (in patients with diabetes mellitus) levels, improving exercise tolerance and quality of life.

The first visit (V0) is an inclusion in the study. During this visit, an attempt to correct or start (if it had not been started before) antiplatelet, hypolipidemic, antihypertensive and antianginal therapy will be made.

The second visit (V1) is planned for each patient three months after the first visit (V0). During the second visit number of patients who reached target levels of BP, LDL-C, frequency of angina attacks will be assessed. If necessary, correction of therapy will also be made.

The third visit (V2) is planned for each patient one year after the first visit (V0). During the third visit reaching target BP, LDL-C levels, frequency of angina attacks will be assessed. If necessary, therapy correction will be recommended.

The last visit - telephone contact with patients - is expected in 2 years after the first visit. During that visit it is planned to assess life status, complications and current medical treatment.

ELIGIBILITY:
Inclusion Criteria:

All patients with documented IHD having consequentially come for the first time for consultation to the specialized cardiology department of the scientific research center from December 31, 2017 to December 31, 2022.

Documented IHD:

1. Positive results of the angina questionnaire (typical angina)
2. Positive exercise electrocardiography or stress echocardiography, plus one of the following criteria:

   * ischemia documented by scintigraphy study
   * invasive coronary angiography data (stenosis of at least 75% in at least one main coronary artery)
   * previous coronary revascularization (percutaneous coronary intervention (PCI), coronary artery bypass graft surgery (CABG))
   * previous myocardial infarction
   * patients who had elective PCI or CABG

Exclusion Criteria:

* Patients with acute IHD (less than 30 days since the last ischemic event with or without invasive procedures for the treatment of the event)
* Patients' refuse to follow the study's graphic of doctors' visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with documented IHD having consequentially come for consultation to the specialized cardiology department of the scientific research center from December 31, 2017 to December 31, 2022
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence to life-modifying treatment | 1 year
  The Adherence scale of the Russian National Society of evidence based pharmacotherapy modified for patients with coronary heart disease will be used to assess patients' adherence to treatment. The patients will be asked questions about taking prescribed medications as recommended by a doctor.
  The score system with the min value in the scale 0 and the max value 4 is used for the assessment of the results: 0 - adherent, 1-2 - partially adherent, 3 - partially non-adherent, 4 - non adherent.
Achievement of the target LDL-C and BP levels | 1 year
  Target LDL-C levels - less than 1.8 mmol/l, target BP levels - less than 140/90 mmHg

SECONDARY OUTCOMES:
all-cause mortality | 2 years
Myocardial Infarction | 2 years
  description - the total number of events
Stroke | 2 years
  description - the total number of events
Unplanned hospitalization for cardiovascular diseases | 2 years
  description - the total number of events
Myocardial revascularization | 2 years
  description - the total number of events
improvement of the functional class of angina in at least 1-grade level | 1 year
  Assessment of the functional class of angina will be made according to the Canadian Cardiovascular Society grading of angina pectoris
Compliance to life-modifying treatment | 1 year
  Necessity of the use of the following drugs will be investigated for each patient: antiplatelets, anticoagulants, hypolipidemic drugs, beta-blockers, ACE-inhibitors/ARBs.
  Later, percent of the drugs that each patient actually takes will be calculated (for example, three drugs are indicated and two are taken - (2/3)*100 = 66.6%).
  In the end, the mean adherence to therapy in the investigated group will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Martsevich, PhD, Study Chair — National Research Center for Preventive Medicine; Ekaterina Zharkova, MD, Principal Investigator — National Research Center for Preventive Medicine
Locations (1):
- National Research Center for Preventive Medicine, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martsevich S.Yu., Zharkova E.D., Kutishenko N.P., Lukina Yu.V., Tolpygina S.N., Voronina V.P., Zagrebelnyy A.V. An Attempt to Accord the Quality of Therapy of Stable Coronary Heart Disease Patients with Current Clinical Guidelines (ALIGN study): Design and the First Results. Rational Pharmacotherapy in Cardiology. 2020;16(1):75-81. (In Russ.) https://doi.org/10.20996/1819-6446-2020-02-08
- [Result] Martsevich S.Y., Lukina Y.V., Zharkova E.D., Kutishenko N.P. Treatment Adherence to Drug Therapyin Patients with Stable Coronary Artery Disease During the COVID-19 Pandemic. Rational Pharmacotherapy in Cardiology. 2021;17(1):99-104. https://doi.org/10.20996/1819-6446-2021-01-06
- [Result] Zharkova E.D., Martsevich S.Yu., Lukina Yu.V., Kutishenko N.P., Drapkina O.M. Assessment of the Quality of Drug Therapy in Patients with Stable Coronary Artery Disease in the Second Stage of the ALIGN Study. Rational Pharmacotherapy in Cardiology. 2022;18(3):306-310. (In Russ.) https://doi.org/10.20996/1819-6446-2022-06-12
- [Result] Zharkova E.D., Martsevich S.Yu., Lukina Yu.V., Kutishenko N.P., Drapkina O.M. The quality of received drug therapy in patients with stable coronary heart disease according to the ALIGN (TherApy in stabLe Coronary Artery dIsease Patients According to Clinical GuideliNes) study. Cardiovascular Therapy and Prevention. 2022;21(9):3371. (In Russ.) https://doi.org/10.15829/1728-8800-2022-3371